CLINICAL TRIAL: NCT05616533
Title: Consistency Evaluation of a Patient-derived Tumor Xenograft Zebrafish Model in Predicting Anti-cancer Efficacy of Conventional Drugs for Gastric Cancer
Brief Title: Evaluation of Consistency of PDX Model for Predicting Therapeutic Effect of Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Hunter Biotechnology Incorporation (Unknown)
Responsible Party: Principal Investigator, Xiaoli JIn, Doctor of Gastrointestinal department of second affiliated hospital of Zhejiang University, Zhejiang University
Other Study IDs: ZRWC_GC_R001
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Precise Prediction of Therapy Efficiency
Keywords: gastric cancer; zebrafish; patient-derived tumor xenograft(PDX) model; prediction; therapy efficiency
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — tumor samples obtained before neoadjuvant treatment and would be transplanted the zebrafish model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- focused group: Advanced gastric patients that will be treated with neoadjuvant therapy are enrolled. Every clinical decision such as regimen or dosage will be decided by their own doctors without any interventions. Tumor samples will be obtained before the first cycle of the treatment and will be transplanted to the zebrafish model. Compared results will be analyzed in future.
  Interventions: Other: biopsy of tumor before treatment

INTERVENTIONS:
Other: biopsy of tumor before treatment — samples obtained from biopsy will be used in the zebrafish PDX model

SUMMARY:
The goal of this study is to compare the tumor response in gastric cancer patients given neoadjuvant chemotherapy with the corresponding result obtained from zebrafish patient-derived tumor xenograft(PDX) model given the same regimen. The main question it aims to answer is whether this PDX model of zebrafish could accurately predict the effect of chemotherapy in advanced gastric cancer. Participants will be given the standard neoadjuvant treatment administrated by their own doctors and tumor response will be observed and recorded. Meanwhile, tumor samples derived from patients before chemotherapy will be transplanted to zebrafish and the same regimen will be given to the PDX models correspondingly. The tumor response data both from clinical practice and PDX model platform will be analysed and compared to evaluate the power of this zebrafish model platform in drug efficiency prediction.

DETAILED DESCRIPTION:
The prognosis of advanced gastric cancer treated with surgery only remains quite disappointed. Adjuvant and neoadjuvant chemotherapy had been greatly raising the survive of advanced gastric cancer. However, how to acquired the tumor sensitivity to the following chemotherapy before the treatment, in order to admit reasonable drugs, avoid unexpected progression of tumor and unnecessary loss of surgical opportunity, remained the focus in this field. Zebrafish CDX/PDX model provides a reliable potential platform for drug sensitivity prediction, but the drug sensitivity result concluded by this platform could not fully represent its actual clinic efficacy in human body. Consistency of therapeutic efficacy could be concluded only by comparing the results both in the human body and the model that was given the same regimens. This is the golden standard to evaluate whether the PDX model of zebrafish could accurately predict the effect of chemotherapy, as well as the primary foundation of the clinical practice with this zebrafish model platform for drug efficiency prediction. Therefore, we intend to carry out this clinical study in gastric cancer patients whom were given neoadjuvant chemotherapy. Enrolled individuals was given a biopsy through endoscopy to obtain samples that would be transplanted to the zebrafish model. Same drugs would be give both for the patient and corresponding zebrafish model, and results would be observed carefully to assess the consistency between the model and the actual practice. This may give strong support for the future clinical use of the platform.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 18-75years,
2. patients with gastric cancer confirmed by histology or cytology at first visit,
3. patients with advanced tumor by imaging evaluation,
4. patients with preoperative neoadjuvant therapy;
5. Eastern Cooperative Oncology Group (ECOG) physical status score of 0 or 1;
6. tolerance to chemotherapy in laboratory examination;
7. hematology examination: no obvious signs of hematological diseases, ANC ≥1.5 × 109/L before enrollment; Platelet count ≥80 × 109/L, HB ≥90 g/L, WBC ≥3.0 × 109/L, and no bleeding tendency;
8. biochemical examination: Total Bilirubin <1.5 times of upper limit of normal value, AST, ALT < 2.5 times of upper limit of normal value, creatinine < 1.5 times of upper limit of normal value;

Exclusion Criteria:

1. patients with inoperable advanced gastric cancer,
2. patients with metastatic or primary gastric cancer,
3. pregnant or lactating women,
4. patients with a history of other malignancies in the last 5 years;
5. for those with a history of uncontrolled epilepsy, central nervous system disease or mental disorders, the severity of the clinical condition was assessed by the investigator as impeding the signing of informed consent or affecting the patient's compliance with oral medication;
6. clinically serious (i.e. active) heart disease, such as symptomatic coronary heart disease, NYHA Class II or more heart failure, or arrhythmias requiring medical intervention; Or a history of myocardial infarction within the last 12 months;
7. severe diabetes-related complications, such as diabetic nephropathy, diabetic ketosis, etc.
8. gastrointestinal obstruction or abnormal physiological function, or malabsorption syndrome, which may affect drug absorption;
9. gastrointestinal bleeding in the last two weeks or at high risk of bleeding as judged by the investigator;
10. patients with known peripheral nerve disease ≥ NCI-CTC AE Grade 1, but only with deep tendon reflexes (DTR) ;
11. organ transplantation requires immunosuppressive therapy;
12. the presence of any active, known or suspected autoimmune disease.
13. uncontrolled severe infection or other severe concomitant disease
14. hypersensitivity to paclitaxel, Oxaliplatin, 5-FU, or any clinically useful anti-gastric cancer agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced gastric cancer that will be treated with neoadjuvant chemotherapy, and surgery will be performed after 2 or 3 cycle of neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The coincidence rate of tumor response obtained from 50 PDX models with clinical real tumor response acquired from corresponding patients received neoadjuvant therapy. | about 3 months (from the first cycle of neoadjuvant therapy to the surgery)
  Drugs used in the zebrafish PDX model are as same as those administrated in the clinical practice with the corresponding patient. Immunofluorescence quantitative detection would be used to evaluate the tumor response in PDX model while RECIST 1.1 and Becker criterion would be applied to evaluate the real tumor response in clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Jin, Dr, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- gastrointestinal department of second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided